CLINICAL TRIAL: NCT04058704
Title: A Multi-center, Prospective Study to Determine the Efficiency of Icotinib Combined With Radiation Therapy Early Intervention or Late Intervention For NSCLC Patients With Brain Metastases and EGFR(Epidermal Growth Factor Receptor) Mutation
Brief Title: A Study to Determine the Efficiency For Brain Metastasis NSCLC Patients Treated With Icotinib Alone or Combined With Radiation Therapy
Acronym: SMART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV99
Record Dates: First submitted 2019-08-11; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases
Keywords: EGFR-TKI; NSCLC; Icotinib; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Experimental): Icotinib is administered orally three times per day. Radiation therapy (SRS/ WBRT/ HA-WBRT/SMART) start in 1 month since take icotinib orally.
  Interventions: Drug: Icotinib; Radiation: SRS/WBRT/HA-WBRT/SMART
- Late intervention (Experimental): Icotinib is administered orally three times per day. Until emerge the progression of the disease, then is given radiation therapy (SRS/WBRT/HA-WBRT/SMART)
  Interventions: Drug: Icotinib; Radiation: SRS/WBRT/HA-WBRT/SMART

INTERVENTIONS:
Drug: Icotinib — 125mg Tid/375mg per day
Radiation: SRS/WBRT/HA-WBRT/SMART — >3 with WBRT/HA-WBRT/SMART or 1-3 with SRS

SUMMARY:
The purpose of this study is to evaluate the efficacy of icotinib alone or in combination with radiation therapy for NSCLC patients harboring EGFR mutation with brain metastases. The primary endpoint is overall survival .

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is one of the malignant tumors with the highest incidence of brain metastases, and most patients died due to the progression of brain metastases. Some research show that icotinib combined with radiation therapy can improve the efficiency of NSCLC with brain metastases, but there is still controversial about the timing of radiation therapy intervention . This study is a prospective, multi-center, randomized, controlled trial of icotinib combined with early intervention or late intervention radiation therapy for NSCLC patients harboring EGFR mutation with brain metastases. They will be treated with icotinib and divided into 2 groups. Group 1: the radiation therapy will start within 1 month after icotinib treatment; Group2: the patients will be treated with icotinib first, radiation therapy intervene if disease progress.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small-cell lung cancer (NSCLC)
* Positive EGFR mutation（Ex19del or 21L858R）
* Primary diagnosis of brain metastases
* Have one or more measurable encephalic lesions according to RECIST
* Extracranial transfer organ≤3
* ECGO:0-2
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.
* Adequate renal function: Serum creatinine ≤1.5 x ULN, or ≥ 50 ml/min.
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and -Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
* Female subjects should not be pregnant.
* All human subjects should able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Written informed consent provided.

Exclusion Criteria:

* Previous usage of EGFR-TKI : gefitinib, erlotinib, icotinib，or any other TKI
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.
* Allergic to Icotinib.
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
* Pregnancy or breast-feeding women.
* Participate in the other anti-tumor clinical trials in 4 weeks. have quit from the trail before.
* Any other serious underlying medical, psychological and other condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from date of randomization until the date of death, assessed up to 36 months.

SECONDARY OUTCOMES:
Progression-free survival of intracranial lesions | from date of randomization until the date of progression, assessed up to 10 months
disease control rate of intracranial lesions | from date of randomization until the date of progression, assessed up to 18 months
Quality of life measured by FACT-L/LCS 4.0 | from date of randomization until the date of death from any cause, assessed up to 36 months
  measured by FACT-L/LCS 4.0
Neurocognitive function changes measured by MMSE | from date of randomization until the date of death from any cause, assessed up to 36 months
  measured by MMSE
Observing acute and late toxicity assessed by CTCAE v4.0 | from date of randomization until the date of death from any cause, assessed up to 36 months
  Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Chen Ming, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China